CLINICAL TRIAL: NCT07042672
Title: Behavioral Therapy With and Without GLP-1 Analogue in Patients With Morbid Obesity and Binge Eating Disorder: A Clinical Prospective Observational Study on Body Weight, Binge Eating Behavior, and Harmful Coping Strategies
Brief Title: Behavioral Therapy and GLP-1 Analogue Effects on Binge Eating, Weight, and Coping in Obesity
Acronym: BETTER-GLP1
Status: Recruiting | Type: Observational
Sponsor: Haukeland University Hospital (Other)
Collaborators: University of Bergen (Other)
Responsible Party: Sponsor
Other Study IDs: 2025-854686
Record Dates: First submitted 2025-04-03; First posted 2025-06-29 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-09

CONDITIONS: Binge Eating Disorder Associated With Obesity; Binge Eating Disorder; Eating Disorder Binge; Eating Disorders; GLP-1; CBT; Obesity &Amp; Overweight
MeSH Terms: conditions — Binge-Eating Disorder; Feeding and Eating Disorders; Obesity; Overweight | interventions — Glucagon-Like Peptide 1

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

GROUPS / COHORTS (2):
- Group-GLP1: Participants receiving standard lifestyle treatment including CBT-E group therapy and individual clinical consultations, in combination with a GLP-1 analogue prescribed by their physician (e.g., liraglutide, semaglutide, or tirzepatide) for weight management. GLP-1 analogue selection, dosage, and duration follow routine clinical practice.
  Interventions: Drug: GLP-1; Behavioral: CBTe Group Therapy
- Group-NoMED: Participants receiving standard lifestyle treatment including CBT-E group therapy and individual clinical consultations, but without use of GLP-1 analogues or other appetite-suppressing medications.
  Interventions: Behavioral: CBTe Group Therapy

INTERVENTIONS:
Drug: GLP-1 — Subcutaneous GLP-1 receptor agonist prescribed for weight management according to routine clinical practice. Acceptable agents include liraglutide (up-titrated to ≤ 3.0 mg daily), semaglutide (≤ 2.4 mg weekly), or tirzepatide (≤ 15 mg weekly). Dose escalation and maintenance follow approved product labels and treating-physician judgment. Planned treatment duration: 12 months or longer.
  Groups: Group-GLP1
Behavioral: CBTe Group Therapy — Ten weekly 2-hour group sessions based on Cognitive Behavioral Therapy-Enhanced (CBT-E) plus individualized lifestyle consultations every 4 months over a 12-month period. Content targets eating patterns, weight-management behaviors, and emotion-regulation skills. Delivered by trained multidisciplinary staff at the Obesity Centre.

SUMMARY:
This study is a clinical, longitudinal, non-randomized, prospective observational study that seeks to compare the treatment effects and safety of using GLP-1 analogues versus not using appetite suppressants during a lifestyle treatment program that includes individual consultations every fourth month and 10 weeks of CBT-E group therapy in patients with both obesity and BED.

The primary objective of this study is to evaluate the impact on BED symptomatology, while the secondary objectives include examining the potential adoption of alternative harmful coping mechanisms. Additionally, the study will assess psychological well-being and weight changes and their consequent influence on obesity-associated comorbid conditions.

Adult patients with coexisting obesity and BED presenting at the Obesity clinic at Haukeland University Hospital, Bergen, Norway, will be included Patients will be divided into two groups: Group-GLP1 (n = 40), who will use GLP-1 analogues, and Group-NoMED (n = 40), who will not use appetite suppressants. Both groups will otherwise follow the routine standardized patient care pathway with follow-up controls every four months and participation in CBT group therapy sessions.

Changes in symptoms of BED, alternative harmful coping strategies and mental health will be recorded at baseline and 12 months using patient-reported questionnaires, as well as anthropometric and biochemical data.

ELIGIBILITY:
Inclusion criteria

1. Severe obesity defined as BMI >40 kg/m2 or 35 kg/m2 with obesity-related comorbidities: coronary artery disease, heart failure, hypertension, atrial fibrillation, cerebral stroke, venous thromboembolism, obstructive sleep apnea, obesity hypoventilation syndrome, type 2 diabetes mellitus, non-alcoholic fatty liver disease, dyslipidemia, osteoarthritis and polecystic ovary syndrome
2. Age between 18 to 65 years
3. Diagnosis of BED according to DSM-5 criteria
4. Willingness to participate and provide informed consent
5. Able to understand and communicate in Norwegian

Exclusion criteria

1. Pregnant or lactating women, as well as women planning pregnancy within one year.
2. Current use medications with major effects on appetite regulation or weight (including, but not limited to systemic glucocorticoids and antipsychotic medication)
3. Renal failure with estimated glomerular filtration rate less than 30 mL/min/1,73m2
4. Liver failure with either ASAT and/or ALAT 5 times upper reference limit, or ALP and/or GT more than 3 times upper reference limit, or clinical signs of liver decompensation
5. Active cancer
6. Previous medullary thyroid cancer
7. Previous pancreatitis
8. Active substance abuse (but previous drug abuse accepted)
9. Medical or psychological treatment within the specialized health care service for eating disorders within the last 6 months.
10. Ongoing severe psychiatric disease that makes them unable to follow the lifestyle treatment program
11. Any illness or prior treatment that in the opinion of the investigator would jeopardize the patient's participation in the study or impact integrity and/or quality of study data.
12. Previous bariatric surgery
13. Use of appetite suppressing drugs (e.g., GLP-1 analogues and/or naltrexone/bupropion) within the last 6 months
14. Participation in another clinical study involving an investigational medicinal product within 1 month prior to study inclusion

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with obesity and binge eating disorder.
  The study will enroll patients with concomitant severe obesity and BED who are referred to the Obesity clinic at Haukeland University Hospital, Norway. All potentially eligible participants will be routinely screened for BED and EDE interview (gold standard) will be used to formally diagnose BED according to the DSM-5.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2025-07-01 (Actual); Primary Completion 2027-11-05 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in EDE-Q Global Score From Baseline to 12 Months | Baseline and 12 months
  The Eating Disorder Examination Questionnaire (EDE-Q, version 6.0) global score is a validated measure of core eating disorder psychopathology, ranging from 0 to 6, with higher scores indicating greater symptom severity.
  The EDE-Q comprises 28 items and assesses cognitive and behavioral symptoms over the past 28 days, including four subscales: restraint, eating concern, shape concern, and weight concern.
  This outcome measures the mean change in global score from baseline to 12-month follow-up, comparing participants receiving GLP-1 analogue treatment (Group-GLP) versus those not receiving appetite suppressants (Group-NoMED).

SECONDARY OUTCOMES:
Proportion of Participants With Increase in Composite Harmful Coping Endpoint (CHCE) From Baseline to 12 Months | Baseline and 12 months
  The Composite Harmful Coping Endpoint (CHCE) captures the emergence of new harmful coping behaviors from baseline to 12-month follow-up. It is defined as a binary outcome, scored as positive if any of the following occur:
  * Deliberate self-harm (DSHI score > 0)
  * Alcohol misuse (AUDIT >= 8 for men, >= 6 for women)
  * Drug misuse (DUDIT > 6 for men, > 2 for women)
  Each of the three components is dichotomized using validated clinical thresholds. Participants with no indication at baseline who cross threshold for any of the three domains at 12 months are considered to have developed a new harmful coping strategy (CHCE = 1). The outcome will compare the proportion of participants with CHCE = 1 between Group-GLP and Group-NoMED.
  DSHI; Deliberate Self-Harm Inventory (range 0-17, higher is worse), AUDIT; Alcohol Use Disorders Identification Test (range 0-40, higher is worse), DUDIT; Drug Use Disorders Identification Test (range 0-44, higher is worse)

OTHER OUTCOMES:
Qualitative Evaluation of Patient Experiences With Combined CBT and GLP-1 Treatment | 12 months
  A subset of study participants (n = 12) receiving GLP-1 analogue treatment will be invited to participate in structured in-depth interviews at 12-month follow-up. Interviews will explore patient experiences related to appetite regulation, eating habits, emotion regulation, and coping strategies during the treatment period. Interviews will be audio-recorded, transcribed, and analyzed using thematic content analysis. This qualitative outcome complements quantitative endpoints by providing insight into subjective treatment experiences.
Mean Difference in Change in AUDIT Score Between Groups From Baseline to 12 Months | From baseline to 12 months
  The Alcohol Use Disorders Identification Test (AUDIT) is a 10-item screening tool developed by the WHO to assess alcohol consumption, drinking behaviors, and alcohol-related problems. Each item is scored from 0 to 4, yielding a total score range of 0 to 40. Higher scores indicate more severe alcohol-related problems.
  This outcome assesses the mean difference in AUDIT score change from baseline to 12-month follow-up between participants receiving GLP-1 analogues (Group-GLP) and those not receiving appetite suppressants (Group-NoMED).
Mean Difference in Change in DUDIT Score Between Groups From Baseline to 12 Months | Baseline and 12 months
  The Drug Use Disorders Identification Test (DUDIT) is an 11-item screening tool for drug misuse, with total scores ranging from 0 to 44. Higher scores indicate greater severity of drug-related problems.
  This outcome assesses the mean difference in DUDIT score change from baseline to 12-month follow-up between participants receiving GLP-1 analogues (Group-GLP) and those not receiving appetite suppressants (Group-NoMED).
Mean Difference in Change in DSHI Score Between Groups From Baseline to 12 Months | Baseline and 12 months
  The Deliberate Self-Harm Inventory (DSHI) is a 17-item self-report questionnaire assessing the presence of specific self-injurious behaviors. Each item is scored 0 (absent) or 1 (present), yielding a total score ranging from 0 to 17. Higher scores reflect a greater number of different self-harm methods.
  This outcome assesses the mean difference in DSHI score change from baseline to 12-month follow-up between participants receiving GLP-1 analogues (Group-GLP) and those not receiving appetite suppressants (Group-NoMED).
Mean Difference in Change in DERS Score Between Groups From Baseline to 12 Months | Baseline and 12 months
  The Difficulties in Emotion Regulation Scale (DERS) is a 36-item self-report questionnaire that assesses emotional dysregulation across six domains, including nonacceptance of emotional responses, difficulties in goal-directed behavior, impulse control difficulties, lack of emotional awareness, limited access to emotion regulation strategies, and lack of emotional clarity. Total scores range from 36 to 180, with higher scores indicating greater emotion regulation difficulties.
  This outcome assesses the mean difference in DERS score change from baseline to 12-month follow-up between participants receiving GLP-1 analogues (Group-GLP) and those not receiving appetite suppressants (Group-NoMED).
Mean Difference in Change in BDI-II Score Between Groups From Baseline to 12 Months | Baseline and 12 months
  The Beck Depression Inventory-II (BDI-II) is a 21-item self-report questionnaire used to assess the severity of depressive symptoms over the past two weeks. Each item is scored from 0 to 3, producing a total score range from 0 to 63. Higher scores indicate more severe depressive symptoms.
  This outcome assesses the mean difference in BDI-II score change from baseline to 12-month follow-up between participants receiving GLP-1 analogues (Group-GLP) and those not receiving appetite suppressants (Group-NoMED).
Mean Difference in Change in BAI Score Between Groups From Baseline to 12 Months | Baseline and 12 months
  The Beck Anxiety Inventory (BAI) is a 21-item self-report questionnaire designed to measure the severity of anxiety symptoms over the past week. Each item is scored from 0 to 3, yielding a total score range from 0 to 63. Higher scores indicate more severe anxiety symptoms.
  This outcome assesses the mean difference in BAI score change from baseline to 12-month follow-up between participants receiving GLP-1 analogues (Group-GLP) and those not receiving appetite suppressants (Group-NoMED).
Mean Difference in Change in CIA Score Between Groups From Baseline to 12 Months | Baseline and 12 months
  The Clinical Impairment Assessment Questionnaire (CIA) is a 16-item self-report measure that assesses psychosocial impairment secondary to eating disorder symptoms over the past 28 days. Total scores range from 0 to 48, with higher scores indicating greater functional impairment.
  This outcome assesses the mean difference in CIA score change from baseline to 12-month follow-up between participants receiving GLP-1 analogues (Group-GLP) and those not receiving appetite suppressants (Group-NoMED).
Mean Difference in Change in Body Weight and BMI Between Groups From Baseline to 12 Months | Baseline and 12 months
  Body weight (in kilograms) and Body Mass Index (BMI, in kg/m²) are measured at baseline and 12-month follow-up.
  Body weight is measured by InBody 770. This outcome assesses the mean difference in change in body weight and BMI between participants receiving GLP-1 analogues (Group-GLP) and those not receiving appetite suppressants (Group-NoMED).
Mean Difference in Change in Systolic and Diastolic Blood Pressure Between Groups From Baseline to 12 Months | Baseline and 12 months
  Systolic and diastolic blood pressure are measured in mmHg using an automated oscillometric device (Welch Allyn) at baseline and 12-month follow-up.
  This outcome assesses the mean difference in change in blood pressure between participants receiving GLP-1 analogues (Group-GLP) and those not receiving appetite suppressants (Group-NoMED).
Mean Difference in Change in Biochemical Markers of Metabolic Disease Between Groups From Baseline to 12 Months | Baseline and 12 months
  Fasting blood samples are analyzed for metabolic markers including high-sensitive C-reactive protein (CRP), hemoglobin A1c (HbA1c), total cholesterol, HDL-cholesterol, LDL-cholesterol, and triglycerides. Values are reported in standard clinical units (e.g., mmol/L or % for HbA1c).
  This outcome assesses the mean difference in change in these biochemical markers from baseline to 12-month follow-up between participants receiving GLP-1 analogues (Group-GLP) and those not receiving appetite suppressants (Group-NoMED).

CONTACTS AND LOCATIONS:
Locations (1):
- Haukeland University Hospital, Bergen, Vestland, Norway

IPD SHARING:
Plan to Share IPD: No